CLINICAL TRIAL: NCT00225810
Title: Multicentre, Controlled, Randomised, Open, Cross-over Study Comparing the Acceptability of Pentasa® Sachets Versus Pentasa® Tbl. 500 mg in Children With Crohn´s Disease
Brief Title: A Study Comparing the Acceptability of Pentasa® Sachets Versus Pentasa® Tablets in Children With Crohn´s Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PENT-IBD-CH CZ
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Crohn's Disease

SUMMARY:
The primary objective of the clinical trial is the assessment of the acceptability of the new Pentasa formulation - PentasaR Sachets in comparison with the reference PentasaR tablets 500 mg in children with Crohn's disease. After the screening period (which includes medical history, physical examination, basic haematology, serum chemistry , urine analysis and stool microbiology , PCD Activity Index )patients will receive (visit I) Pentasa sachets 1g or Pentasa tablets 500mg for next 4 weeks according to the randomisation scheme in common dose 2× 1 g of PentasaR Sachets 1 g or PentasaR tablets 500 mg. The formulation of Pentasa will be switched at Visit 2, patients will receive the medication for next 4 weeks. Patients will record the acceptability of the both forms of the medication.

In 6 patients from each group (selected by the randomization), stool and urine will be taken to assess concentrations of mesalazine and N-acetylmesalazine during Visit 2 and Visit 3. Adverse events will be recorded during the whole course of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnose of Crohn's disease
* Age 8-18 years, both sexes
* Weight above 40 kg
* Oral maintenance treatment with 5-ASA and any concomitant antinflammatory medication (maintained at the same dose during the study) before inclusion is permitted,
* written informed consent obtained (patient and his/her guardian)

Exclusion Criteria:

* Patients with a history of allergy to salicylates
* Patients with known significant hepatic or renal function abnormalities
* Positive enteric pathogens in stool (Salmonella, Shigella, Yersinia, Campylobacter)
* Pregnant or lactating women
* Patients with a known history of disease, including mental/emotional disorder, that would interfere with their participation in the study,
* Patients who participated in another clinical study in the last 3 months,
* Patients who are unable to comply with the requirements of the protocol
* Patients who are unable to fill in the diary cards

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2005-10; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To assess the acceptability of Pentasa Sachets in comparison with the reference Pentasa tablets 500mg in children with Cohn's disease.

SECONDARY OUTCOMES:
To compare the safety of both formulations of Pentasa.
To compare the concentration of mesalazine and N-acetylmesalazine in urine and stool during the administration of both formulations of Pentasa.
To compare the PCD activity index at Week 4 and 8 Phase IV Study design: instead of Single Blind use Open Total enrollment: 29 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (2):
- Czechia (2):
  - Faculty Hospital Bulovka, Paediatric Clinic, Prague
  - Faculty Hospital Motol, Paediatric Clinic, Prague